CLINICAL TRIAL: NCT06259279
Title: High Impact Training to Patients with Prostate Cancer and Bone Metastases
Acronym: HIP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Copenhagen University Hospital at Herlev (Other)
Responsible Party: Principal Investigator, Anne-Mette Ragle, Principal Investigator, Copenhagen University Hospital at Herlev
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: AMRagle
Record Dates: First submitted 2024-01-29; First posted 2024-02-14 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Prostate Cancer
Keywords: bone metastases; exercise; bone mineral density; resistance and impact training; antitumor immunity
MeSH Terms: conditions — Prostatic Neoplasms; Motor Activity

STUDY DESIGN:
Intervention Model Description: RCT
Who Masked: Outcomes Assessor
Masking Description: Testers of physical tests (Handgrip strength test and chair-stand-test) and the the statistician will be blinded for allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention Group (Experimental): Patients in the intervention group will receive a 32-week exercise-based intervention that includes supervised and group-based exercise training in the hospital, twice a week. Each session lasts approximately 30 minutes.
  Interventions: Behavioral: High intensity high impact exercise intervention
- Control Group (No Intervention): standard care. Patients in the control group are referred to the municipal standard rehabilitation programs if the patient so wishes.

INTERVENTIONS:
Behavioral: High intensity high impact exercise intervention — Patients in the intervention group will receive a 32-week exercise-based intervention that includes:
  - Supervised and group-based exercise training in the hospital, twice a week. Each session lasts approximately 30 minutes.
  Arms: Intervention Group

SUMMARY:
HIP is a randomized controlled trial. The aim is investigate the effect, safety and feasibility of brief, high-impact exercise targeting bones in patients with prostate cancer and bone metastases. Furthermore, to investigate the effects of the intervention on bone status (bone mineral density) and body composition, physical function and performance, patient reported quality-of-life outcomes, falls and hospitalizations. The effects of resistance training on the antitumor immunity will be assessed in the peripheral blood and tumor biopsies (HIPimmune).

DETAILED DESCRIPTION:
Participants assigned to the intervention group will participate in a 32-week, twice-weekly, 30-minute, supervised HIP program at the hospital in Herlev, Denmark. To ensure a safe transition to high-intensity exercise, the first eight weeks of the intervention includes self-bodyweight and low-impact variations with a focus on getting used to use weight training equipment and gradually learning the movement patterns of the HIP exercises. All participants should be able to perform the four basic exercises of the intervention within two months. The resistance exercises (deadlift, overhead press, and squats) will be performed in five sets of five repetitions for the remaining intervention period, maintaining an intensity of > 80% to 85% of 1 repetition maximum (RM). Blood samples and tumor biopsies will be taken at different timepoints of the exercise intervention (HIPimmune) and analyzed for lymphocyte entitumor responses.

ELIGIBILITY:
Inclusion Criteria:

* Patients with metastatic hormone sensitive prostate cancer (mHSPC)
* Patients must have bone metastases according to the most recent imaging (Bone scan, CT, MRI and/or PET)
* Patients must be treated with androgen deprivation therapy (ADT) (orchiectomy, luteinizing hormone-releasing hormone (LHRH) agonist or antagonist treatment) started < 12 months ago. Additional treatment in the mHSPC setting, i.e., radiotherapy (RT) of the prostate, novel hormone agents (NHA) and/or docetaxel is permitted
* Patients must have an Eastern Cooperative Oncology Group (ECOG) performance status score <2
* Patients must be able to speak and read Danish and provide a signed informed consent form
* Patients must be ambulatory without walking aids

Exclusion Criteria:

* Patients with any physical condition that interferes with the performance of physical exercise training
* Patients with presence of any musculoskeletal, cardiovascular, or neurologic conditions that may prevent patients from exercising
* Patients with bone pain requiring opioids
* Patients with planned or prior palliative radiation therapy to the bone
* Patients with major surgery within the past 6 months

HIPimmune: all patients included in HIP are eligible for HIPimmune

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Estimated)
Dates: Start 2024-02-06 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Lower body strength measured with the 30-second chair stand test (30s-CST) | baseline, 16 weeks, 32 weeks and 44 weeks
  Number of stands a participant can complete in 30-seconds from a seated position with their arms crossed over the chest. The assesment will be conducted by blinded physiotherapist

SECONDARY OUTCOMES:
Fat free mass (kg) | Change measures baseline, 32 weeks
  Measured with DXA scans
Body fat (% and kg) | Change measures baseline, 32 weeks
  Measured with DXA scans
Whole Body (BMC, g) | Change measures baseline, 32 weeks
  Measured with DXA scans
Whole Body (BMD, g/cm2) | Change measures baseline, 32 weeks
  Measured with DXA scans
Whole body T-score | Change measures baseline, 32 weeks
  Measured with DXA scans
Lumbar spine (L1-L4 BMD, g/cm2) | Change measures baseline, 32 weeks
  Measured with DXA scans
Lumbar spine T-score | Change measures baseline, 32 weeks
  Measured with DXA scans
Total Hip BMD, g/cm2 | Change measures baseline, 32 weeks
  Measured with DXA scans
Total hip T-score Os Calcis BMD, g/cm2 Os calcis T-score | Change measures baseline, 32 weeks
  Measured with DXA scans
Total hip T-score | Change measures baseline, 32 weeks
  Measured with DXA scans
Os Calcis BMD, g/cm2 | Change measures baseline, 32 weeks
  Measured with DXA scans
Os calcis T-score | Change measures baseline, 32 weeks
  Measured with DXA scans
Handgrip strength | baseline, 16 weeks, 32 weeks and 44 weeks
  Handgrip strength grip test, (measured in Kg, higher score is better outcome)
Quality of life (QOL) | Change measures baseline, 16 weeks, 32 weeks and 44 weeks
  Measured with the Functional Assessment of Cancer Therapy-Prostate. the questionnaire is divided into several sub-topics, and it differs from topic to topic whether a high score is best. Minimum score:0 and maximum score 4
Fatigue | Change measures baseline, 16 weeks, 32 weeks and 44 weeks
  Measured with the Functional Assessment of Chronic Illness Therapy - Fatigue Scale. Low score is a better outcome the minimum score is 0, maximum score is 4
Safety (adverse events) | Through study completion, an average of 1 year
  Safety is measured by registration of bone fracture grade > 2 according to Common Terminology Criteria for Adverse Events (CTCAE) grading criteria. Adverse events as musculoskeletal grade > 2 including pain, or cardiac disorders according to CTCAE, and sprains requiring medical treatment.
  Grade 1 Mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated. Grade 2 Moderate; minimal, local or noninvasive intervention indicated; limiting age, appropriate instrumental ADL*. Grade 3 Severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self care ADL**. Grade 4 Life-threatening consequences; urgent intervention indicated. Grade 5 Death related to AE.
Hospitalizations | Through study completion, an average of 1 year
  Registration of hospital admissions in number
Hospitalizations, causes | Through study completion, an average of 1 year
  Registration of causes for hospital admissions
Hospitalizations, length of hospitalizations | Through study completion, an average of 1 year
  Registration of hospital admissions in days
Falls | Through study completion, an average of 1 year
  Participants will be asked to report incidence of any falls in the project period . Falls requiring treatment will be registered as adverse events and be reported according to CTCAE.
Feasibility measured by dropout | Through study completion, an average of 1 year
  Feasibility is assessed by dropout in the study
Feasibility measured by recruitment | Through study completion, an average of 1 year
  Feasibility is assessed by recruitment, numbers of included patients compared to number of eligible patients
Feasibility measured by adherence. | Through study completion, an average of 1 year
  Feasibility is assessed by adherence. How many times the patients participate in the execise sessions . Numbers from 0-64. Higher score is better.
Physical activity | Change measures baseline, 16 weeks, 32 weeks and 44 weeks
  Data of daily physical activity will be assessed in the intervention period using the Physical Activity Scale 2 (PAS -2), which measure physical activity levels
Qualitative assessment of patients' experiences | Up to 6 months after study completion
  Qualitative individual semi-structured interviews with participants from the intervention group
HIPimmune: Immune response in peripheral blood and tumor | Baseline, week 8, week 32, week 44
  Flow-cytometric analysis of circulating immune cell frequencies (T, B, NK cells and myeloid cells) longitudinally during the study period, both before and after the exercise intervention (in the intervention arm). Additionally, prostate biopsies around week 32 will be stained by immunohistochemistry for infiltrating immune cells (T and NK cells).

CONTACTS AND LOCATIONS:
Overall Officials: Anne-Mette Ragle, PhD student, Principal Investigator — Copenhagen University Hospital at Herlev; Peter B Østergren, Study Director — Peter Østergren; Katharina Leuchte, Dr. med., Study Director — University Hospital Copenhagen Herlev, National Center for Cancer Immune Therapy (CCIT)
Locations (1):
- Herlev and Gentofte Hospital, Herlev, Herlev, Denmark

REFERENCES:
- [Derived] Ragle AM, Mikkelsen MK, Vinther A, Zerahn B, Bogh Juhl C, Theile S, Madsen K, Nielsen DL, Ostergren PB. High-intensity resistance and impact training for patients with hormone-sensitive prostate cancer and bone metastases-study protocol of a randomized clinical trial. Trials. 2025 Jul 28;26(1):259. doi: 10.1186/s13063-025-08937-0. PMID 40722114